CLINICAL TRIAL: NCT04143139
Title: Assessment of Bone Mineral Density, Vitamin D Status and Calcium Intakes in Ileostomy Patients.
Brief Title: Ileostomy Observation Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Ulster (Other)
Collaborators: University of Naples (Other)
Responsible Party: Sponsor
Other Study IDs: 16/NI/0267
Record Dates: First submitted 2019-10-07; First posted 2019-10-29 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Ileostomy - Stoma
Keywords: Bone mineral density; Ileostomists; Vitamin D; Observational study; Calcium; Phytochemical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Ileal fluid Blood samples - plasma, serum, whole blood, red cells and buffy coat retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD) which is associated with low bone mineral density is divided into 2 major disease entities: Crohn's disease and ulcerative colitis. Medical therapy is directed at controlling symptoms and reducing the underlying inflammatory process. Studies have reported that 60% of patients with Crohn's disease and 15%-30% of patients with ulcerative colitis require surgical intervention for the management of their disease. In the United Kingdom almost 13,000 ileostomy procedures are undertaken annually. A 29.4% prevalence of low bone mineral density (BMD) was reported in a cohort of US patients with IBD and ileostomy who were >5 years postoperative. Possible risk factors for bone loss in patients with IBD and ileostomy are considered to include malabsorption secondary to bowel resection, malnutrition and more aggressive disease and inflammation which led to bowel resection in the first place . These factors also contribute to reduced intestinal absorption of nutrients and vitamins including B & D subsequently leading to potential health complications including low BMI and low lean body mass. It has been reported that IBD patients who have surgical intervention to create ileal pouches also have low levels of vitamin D.

Surgical procedures such as an ileostomy alter the normal anatomy and physiology of the small intestine. Bile acid (BA) malabsorption which is common to IBD is caused by impaired conjugated BA reabsorption and a consequence, numerous pathological sequelae may occur, including the malfunction of lipid digestion . Further, bacterial overgrowth can lead to deconjugation of bile salts, leading to formation of free bile acids, again inducing dietary fat malabsorption, which in turn can lead to vitamin D deficiency. As vitamin D is a fat-soluble vitamin, malfunction of lipid digestion or absorption is problematic.

Given the paucity of data in the area of ileostomy patients BMD, vitamin D status and calcium intake, we will establish baseline observations within the Northern Ireland (NI) population with an observational study to assess bone mineral density (Dexa), collecting ileal fluid and plasma samples assessing vitamin D status, calcium, dietary intake and other measures including questionnaires on quality of life and exercise.

ELIGIBILITY:
Inclusion Criteria:

* undergone an ileostomy and be more than 2 year post-operative
* non smoking

Exclusion Criteria:

* not undergone an ileostomy and/or is less than 2 year post-operative
* smoker.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ileostomy patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Bone Density | 1 day, 1 measurement
  Dual Energy X-ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
Total serum 25-hydroxyvitamin D [25(OH)D] commercial kit) | 1 day, 1 measurement
  Liquid Chromatography / Mass Spec (LC/MS)
Parathyroid hormone concentrations commercial kit) | 1 day, 1 measurement
  Commercial kit
Serum adjusted calcium | 1 day, 1 measurement
  Commercial kit
Lipid profile | 1 day, 1 measurement
  Commercial kit
Plasma glucose | 1 day, 1 measurement
  Commercial kit
Dietary intake, | 1 day, 1 measurement
  Food dairy and Vitamin D Food Frequency Questionaire
Phytochemical concentrations (plasma and ileal fluid) analysis | 1 day, 1 measurement
  Gas Chromatography Mass Spect (GCMS) and Liquid Chromatography / Mass Spec (LC/MS) Mass Spec (LC/MS)
Quality of life (QoL) questionnaire | 1 day, 1 measurement
  Coloplast Stoma-QoL; 20 questions, 4-point scale. Higher value representing higher QoL
Heath and well being questionnaire | 1 day, 1 measurement
  SF36v2, Higher value representing a greater health and well-being status.
Recent Physical Activity Questionnaire (RPAQ) | 1 day, 1 measurement
  Validated questionnaire measuring time spent in active and sedentary behaviour.
Dietary component (plasma and ileal fluid) concentrations such as polyunsaturated fatty acids, endocannabinoids | 1 day, 1 measurement
  Gas Chromatography Mass Spect (GCMS) and Liquid Chromatography / Mass Spec

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tagliamonte S, Gill CIR, Pourshahidi LK, Slevin MM, Price RK, Ferracane R, Lawther R, O'Connor G, Vitaglione P. Endocannabinoids, endocannabinoid-like molecules and their precursors in human small intestinal lumen and plasma: does diet affect them? Eur J Nutr. 2021 Jun;60(4):2203-2215. doi: 10.1007/s00394-020-02398-8. Epub 2020 Oct 26. PMID 33104865